CLINICAL TRIAL: NCT03338205
Title: The Role of Ketamine as an Adjuvant Therapy for Children With Acute Status Asthmaticus in Pediatric Emergency Medicine Patients: A Pilot Study
Brief Title: The Role of Ketamine as an Adjuvant Therapy for Children With Acute Status Asthmaticus
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to enroll patients
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 51152
Record Dates: First submitted 2017-11-01; First posted 2017-11-09 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Status Asthmaticus
Keywords: ketamine; pediatric status asthmaticus
MeSH Terms: conditions — Status Asthmaticus | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine Treatment (Experimental): Everyone enrolled in study presenting in status asthmaticus to pediatric emergency department at Augusta University will receive a ketamine treatment, who include:
  * Patients with a Clinical Asthma SCore (CAS) of greater than or equal to 10 on presentation and have received at least two (appropriately dosed based on weight) albuterol treatments prior to arrival
  OR
  * Patients with a CAS of ≥ greater than or equal to 10 that have not received treatment prior to arrival and after receiving 1 hour of treatment per the severe asthma pathway do not have a decrease in CAS of greater than 2
  OR
  * Patients with a CAS above > 6 but less than < 10 when as measured 1 hour after initiation of standard treatment per Augusta University's moderate asthma pathway
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 1 mg/kg ketamine bolus IV

SUMMARY:
The purpose of this investigation is to perform a pilot study assessing the safety and utility of intravenous ketamine as an adjuvant therapy in the emergency department setting for pediatric patients in acute status asthmaticus who have failed standard emergency therapy.

DETAILED DESCRIPTION:
This is a pilot study of a cohort of 20 subjects to assess the feasibility, safety and efficacy of ketamine in status asthmaticus.

The study will take place at the Augusta University's pediatric emergency department 24 hours a day. The attending physician who is clinically treating the patient will identify the patient as a potential study candidate (see inclusion criteria). Study team members will then be notified and obtain informed consent for potential participants who meet the inclusion/exclusion criteria.

Once a patient in the Augusta University Children's Hospital of Georgia Pediatric Emergency Department is deemed a potential study subject, informed consent will be obtained by the research study team members. The patient and their parents will be provided with all the required information about the study including potential risks and benefits associated with participation. The information will be presented in a private setting in a language the patient understands. The patient and/or their parent/guardian will have opportunities to ask questions and will be given enough time to consider participation before providing consent. A document will be given to obtain assent/consent that reiterates all the information about the study (including reason for the study, risks, benefits, etc.)

Study team members that will be actively involved in the study will be either pediatric emergency medicine faculty or pediatric emergency medicine fellows that are on staff.

Patients that meet the inclusion and exclusion criteria will have ketamine 1 mg/kg IV bolus administered once informed consent has been obtained.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (≥2 years and ≤ 18 years old)

Patients presenting in status asthmaticus:

* Patients with a CAS of greater than or equal to 10 on presentation that have received at least two (appropriately dosed based on weight) albuterol treatments prior to arrival

OR

* Patients with a CAS of greater than or equal to 10 that have not received treatment prior to arrival and after 1 hour of treatment per the severe asthma pathway do not have a decrease in CAS of greater than 2

OR

* Patients with a CAS above 6 but less than 10 as measured 1 hour after initiation of standard treatment per AU's moderate asthma pathway

Exclusion Criteria:

* Pregnancy
* Congestive Heart Failure or prior diagnosis of cardiovascular disease (congenital or acquired)
* Chronic lung disease outside of a previous diagnosis of Asthma
* Seizure disorder
* Liver disease
* History of hypertension greater than 95% for age
* Obstructive Sleep Apnea with AHI greater than 5
* History of allergic or serious reaction to Ketamine
* Significant history of psychiatric illness defined as any patient with a diagnosis of psychiatric illness meeting the Diagnostic and Statistical Manual of Mental Disorders V criteria (severe Autism)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of ketamine in status asthmaticus by assessing change in clinical asthma score (CAS) | prior to intervention, 30 minutes and 60 minutes after administration of ketamine
  CAS will be documented on admission, prior to intervention, 30 minutes and 60 minutes after administration of ketamine. The CAS is a scoring system to assess the severity of asthma used by Augusta University and is based on physiological measurements and clinical appearance.